CLINICAL TRIAL: NCT01270074
Title: A Phase 3 Multi-centre Randomised Placebo-controlled Study of Azithromycin in the Primary Prevention of Radiologically-defined Bronchiectasis in Infants With Cystic Fibrosis.
Brief Title: Prevention of Bronchiectasis in Infants With Cystic Fibrosis
Acronym: COMBATCF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Queensland (Other)
Collaborators: Telethon Kids Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AZI001; STICK10K0 (Other Grant/Funding Number: Cystif Fibrosis Foundation Therapeutics, INc.)
Record Dates: First submitted 2010-12-23; First posted 2011-01-05 (Estimated); Last update posted 2021-09-16 (Actual); Status verified 2019-11

CONDITIONS: Cystic Fibrosis; Bronchiectasis
Keywords: double blind placebo controlled randomised clinical trial; azithromycin; infant; pediatric; cystic fibrosis; bronchiectasis
MeSH Terms: conditions — Cystic Fibrosis; Bronchiectasis | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- azithromycin liquid preparation (Experimental): azithromycin will be given at a dose of 10mg/kg given three times per week from three months of age to three years of age
  Interventions: Drug: Azithromycin
- inert liquid preparation (Active Comparator): inert liquid preparation will be given three times per week from three months of age to three years of age
  Interventions: Drug: Placebo control

INTERVENTIONS:
Drug: Azithromycin — azithromycin will be given as a liquid preparation at a dose of 10 mg/kg three times per week from three months of age until three years of age
  Other Names: Zithromax
  Arms: azithromycin liquid preparation
Drug: Placebo control — inert liquid preparation will be given three times per week from three months of age to three years of age
  Arms: inert liquid preparation

SUMMARY:
The general aim of this project is to conduct a randomized, double-blind, placebo-controlled clinical trial of azithromycin to determine whether treatment from infancy is safe and will prevent the onset of bronchiectasis. One hundred and thirty infants will be recruited from CF clinics in Australia and New Zealand and treated from 3 months to three years of age. The primary outcome will be the proportion with radiologically-defined bronchiectasis at 3 years of age. Safety and mechanistic evaluations will also be undertaken.

DETAILED DESCRIPTION:
SYNOPSIS OF PROTOCOL

Title Multi-centre randomized placebo-controlled study of azithromycin in the primary prevention of radiologically-defined bronchiectasis in infants with Cystic Fibrosis

Clinical Phase Phase 3

Protocol Number: AZI001

TGA Reference Number:

Protocol Co-Chairs: Peter D. Sly & Stephen M. Stick Microbiology Consultant: Lisa Saiman CT Consultant: Harm Tiddens Statistical Consultant: Robert S Ware

Study Design Randomized, double-blind parallel groups. Participants will be randomized into one of the following 2 groups on a 1:1 ratio with 65 participants per group;

Group A: 10 mg/kg (as 200mg/5ml) azithromycin three times weekly for three years added to standard CF therapy.

Group B: matched placebo three times weekly for three years added to standard CF therapy.

Accrual Objective 130 children

Accrual Period 24 months

Study Duration 36 months

Countries: Australia and New Zealand

Sites: Brisbane Au, Sydney, Au, Melbourne Au, Adelaide Au, Perth Au,Auckland Nz, Christchurch Nz.

Primary Endpoint The primary endpoints are the proportion of children with radiologically-defined bronchiectasis at age 3 years, and the proportion of lung tissue affected by disease at age 3 years.

Secondary Endpoints

* The extent and severity of bronchiectasis at age 3 years
* The volume of trapped gas at age 3 years
* CF-related quality of life
* Time to first pulmonary exacerbation
* Proportion of participants experiencing a pulmonary exacerbation
* Number of courses of inhaled or oral antibiotics
* Number of days of inhaled antibiotics
* Incidence of hospitalizations/Accident and Emergency department (A&E) visits for an acute respiratory exacerbation
* Number of days hospitalized for an acute respiratory exacerbation
* Number of days if intravenous antibiotics
* Body mass index at 3 years of age.

Exploratory Endpoints

* Markers of neutrophilic inflammation
* Markers of oxidative stress
* Composition of airway flora

Safety Endpoints

* Proportion of participants growing P. aeruginosa in BAL
* Age of acquisition of P. aeruginosa in BAL
* Emergence of macrolide-resistant S. aureus, small colony variant S. aureus and non-tuberculous mycobacteria (NTM)
* Treatment-related adverse events
* Haematology and clinical chemistry

Inclusion Criteria Participants who meet all of the following criteria are eligible for enrolment as study participants:

1. Children of either sex with a diagnosis of CF following detection via New Born Screening (NBS) for cystic fibrosis
2. Participants who, in the opinion of the Investigator, are able to comply with the protocol for its duration
3. Written informed consent signed and dated by parent/legal guardian according to local regulations

Exclusion Criteria Participants who meet any of these criteria are not eligible for enrolment as trial participants:

1. Born <30 weeks gestation
2. Prolonged mechanical ventilation in the first 3 months of life
3. Participation in another randomized controlled trial within the 3 months preceding inclusion in this study
4. A significant medical disease or condition other than CF that is likely to interfere with the child's ability to complete the entire protocol
5. Previous major surgery except for meconium ileus
6. Macrolide hypersensitivity

Treatment Description ZITHROMAX® (azithromycin)

Study Procedures The study participants will be stratified by investigational site and randomly assigned to either azithromycin or placebo for three years.

Statistical Considerations Participants will be randomized in blocks to the treatment group or the placebo group using a one-to-one ratio. Randomization will be stratified by study site. This will ensure an approximately equal allocation to each group within each site.

Interim Analyses Interim analyses will occur when the first 50% of children (n=33 per group have completed the 12 month CT and when all subjects have completed the 12 month CT. Interim analyses will determine safety or success (unethical to continue).

Stopping Rules Study enrolment may be stopped if any of the following events occur:

* Death of a participant that is related to study treatment.
* The trial meets the definition of futility or success at either of the planned interim analyses

ELIGIBILITY:
Inclusion Criteria:

1. Children of either sex with a diagnosis of CF following detection via New Born Screening (NBS) for cystic fibrosis
2. Participants who, in the opinion of the Investigator, are able to comply with the protocol for its duration
3. Written informed consent signed and dated by parent/legal guardian according to local regulations

Exclusion Criteria:

1. Born <30 weeks gestation
2. Prolonged mechanical ventilation in the first 3 months of life
3. Participation in another randomized controlled trial within the 3 months preceding inclusion in this study
4. A significant medical disease or condition other than CF that is likely to interfere with the child's ability to complete the entire protocol
5. Previous major surgery except for meconium ileus
6. Macrolide hypersensitivity

Ages: 6 Weeks to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 130 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Proportion of children with radiologically-defined bronchiectasis | at three years of age
  bronchiectasis will be determined from a low dose volumetric chest computed tomography scan performed at 3 years of age
The proportion of lung tissue affected by disease | at three years of age
  Percentage of diseased lung will be determined from a low dose volumetric chest computed tomography scan performed at 3 years of age

SECONDARY OUTCOMES:
extent and severity of bronchiectasis | at three years of age
  bronchiectasis will be determined from a low dose volumetric chest computed tomography scan performed at 3 years of age
CF-related quality of life | at three years of age
  Quality of life questionnaire to be measured at 3 years
time to first pulmonary exacerbation | over the first three years of life
  pulmonary exacerbation will be defined using a standardized instrument
proportion of participants experiencing a pulmonary exacerbation | over the first three years of life
  pulmonary exacerbation will be defined using a standardized instrument
body mass index | at three years of age
  body mass index will be calcualted from hieight and weight measurements taken at 3 years of age.
Proportion of participants growing Pseudomonas aeruginosa in bronchoalveolar lavage | over the first three years of life
  bronchoalveolar lavage will be performed at 3 months, 1 year and 3 years of age
age of acquisition of Pseudomonas aeruginosa | over the first three years of life
Emergence of macrolide-resistant Staphylococcus aureus, small colony variant Staphylococcal aureus and non-tuberculous mycobacterium | over the first three years of life
Volume of trapped gas at age 3 years | at 3 years
  air trapping will be determined from a low dose volumetric chest computed tomography scan performed at 3 years of age

CONTACTS AND LOCATIONS:
Overall Officials: Peter D Sly, MMBS MD DSc, Study Chair — The University of Queensland; Stephen M Stick, MBBChir PhD, Study Chair — Telethon Kids Institute
Locations (10):
- Australia (9):
  - Sydney Children's Hospital, Sydney, New South Wales
  - Westmead Children's Hospital, Sydney, New South Wales
  - Queensland Children's Hospital, Brisbane, Queensland
  - Mater Children's Hospital, Brisbane, Queensland
  - Royal Children's Hospital, Brisbane, Queensland
  - Women's and Children's Hospital, Adelaide, South Australia
  - Monash Medical Centre, Melbourne, Victoria
  - Royal Children's Hospital, Melbourne, Victoria
  - Perth Children's Hospital, Perth, Western Australia
- Starship Hospital, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR

REFERENCES:
- [Background] Douglas TA, Brennan S, Gard S, Berry L, Gangell C, Stick SM, Clements BS, Sly PD. Acquisition and eradication of P. aeruginosa in young children with cystic fibrosis. Eur Respir J. 2009 Feb;33(2):305-11. doi: 10.1183/09031936.00043108. Epub 2008 Nov 14. PMID 19010992
- [Background] Sly PD, Brennan S, Gangell C, de Klerk N, Murray C, Mott L, Stick SM, Robinson PJ, Robertson CF, Ranganathan SC; Australian Respiratory Early Surveillance Team for Cystic Fibrosis (AREST-CF). Lung disease at diagnosis in infants with cystic fibrosis detected by newborn screening. Am J Respir Crit Care Med. 2009 Jul 15;180(2):146-52. doi: 10.1164/rccm.200901-0069OC. Epub 2009 Apr 16. PMID 19372250
- [Background] Stick SM, Brennan S, Murray C, Douglas T, von Ungern-Sternberg BS, Garratt LW, Gangell CL, De Klerk N, Linnane B, Ranganathan S, Robinson P, Robertson C, Sly PD; Australian Respiratory Early Surveillance Team for Cystic Fibrosis (AREST CF). Bronchiectasis in infants and preschool children diagnosed with cystic fibrosis after newborn screening. J Pediatr. 2009 Nov;155(5):623-8.e1. doi: 10.1016/j.jpeds.2009.05.005. Epub 2009 Jul 19. PMID 19616787
- [Derived] Stick SM, Foti A, Ware RS, Tiddens HAWM, Clements BS, Armstrong DS, Selvadurai H, Tai A, Cooper PJ, Byrnes CA, Belessis Y, Wainwright C, Jaffe A, Robinson P, Saiman L, Sly PD; COMBAT CF Study Group. The effect of azithromycin on structural lung disease in infants with cystic fibrosis (COMBAT CF): a phase 3, randomised, double-blind, placebo-controlled clinical trial. Lancet Respir Med. 2022 Aug;10(8):776-784. doi: 10.1016/S2213-2600(22)00165-5. Epub 2022 Jun 2. PMID 35662406
- See also: The Australia Respiratory Early Surveillance Team for Cystic Fibrosis — http://arestcf.org
- See also: Telethon Institute for Child Health Research — http://ichr.uwa.edu.au